CLINICAL TRIAL: NCT02502890
Title: Mechanisms Underlying Asthma Exacerbations Prevented and Persistent With Immune-Based Therapy: A Systems Approach Phase 1 (ICAC-29)
Brief Title: Mechanisms Underlying Asthma Exacerbations Prevented and Persistent With Immune-Based Therapy
Acronym: MUPPITS-1
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT ICAC-29
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Asthma
Keywords: asthma; nested case-control study; difficult-to-control asthma; asthma exacerbations; cold symptoms; gene expression
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Nasal Samples.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Asthma is a growing problem, especially in children. It causes frequent wheezing, shortness of breath, chest tightness, and cough. A cold that is caused by a virus (viral cold) can sometimes make asthma symptoms worse. This study will help investigators learn about the way colds are related to asthma attacks among children who need higher amounts of medications to control their asthma. Investigators want to learn why viral colds sometimes cause asthma attacks and other times do not by studying the immune system response in samples taken from the nose and blood.

DETAILED DESCRIPTION:
This study is a prospective, longitudinal, nested case-control study designed to identify changes in gene transcription predictive of and associated with asthma exacerbations in children ages 6 to 17 years with difficult-to-control, exacerbation-prone asthma.

Participants will be followed prospectively for the onset of a cold and a subsequent asthma exacerbation. An internet-based asthma and cold symptom diary will be accessed by participants using a hand-held device. When the participant reports development of a cold, a clinic visit will be scheduled as soon as possible (within 48 hours of cold symptom onset) to collect blood and nasal samples. A second clinic visit will occur 4-6 days from the onset of cold symptoms to obtain samples after the initial cold, but prior to the use of systemic corticosteroids. Participants will be followed for up to two colds or approximately 6 months after Visit 0, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

Participant(s) who meet all of the following criteria are eligible for enrollment. Participant(s) may be reassessed if not initially eligible. Participants are eligible if they:

* Have a primary place of residence in one of the pre-selected recruitment census tracts as outlined in the Inner City Asthma Consortium (ICAC) Manual of Procedures (MOP);
* Have a diagnosis of asthma made by a clinician >1 year prior to recruitment;
* Have had at least 2 asthma exacerbations in the prior year, defined as a requirement for systemic corticosteroids and/or hospitalization;
* Have the following requirement for asthma controller medication at the Screening and Enrollment Visit (Visit 0) according to the MEDS program[4, 2]:

  * For participants aged 6 to 11 years, treatment with at least fluticasone 250 mcg 1 puff twice daily or its equivalent;
  * For participants ages12 years and older, treatment with at least Advair 250/50 mcg 1 puff twice daily or its equivalent.
* Have peripheral blood eosinophils >=150 per mm^3. Results can be obtained from participation in a previous ICAC study if obtained within 6 months of the Screening and Enrollment Visit (Visit 0);
* Currently a non-smoker;
* Parent/legal guardian is willing to sign the written informed consent;
* Participant is willing to sign the assent form as per central Institutional Review Board (IRB) guidelines;
* Has some form of insurance that covers costs of usual care asthma control and rescue medications at the Screening and Enrollment Visit (Visit 0).

Exclusion Criteria:

Participant(s) who meet any of the following criteria are not eligible for enrollment but may be reassessed. Participant(s) are ineligible if they:

* Are currently pregnant or lactating;
* Are currently receiving treatment with anti-immunoglobulin E (anti-IgE) therapy or have had anti-IgE therapy in the previous 3 months prior to screening;
* Are currently receiving immunotherapy;
* Have clinically significant abnormalities on complete blood count (CBC) with differential as determined by the site study clinician. Results can be obtained from participation in a previous ICAC study [including Registry for Asthma Characterization and Recruitment 2 (RACR2), NCT02513264} if obtained within the last 6 months of Visit 0;
* Was treated with systemic corticosteroids for any medical condition including an asthma exacerbation within the 2 weeks prior to Visit 0;
* Have had a cold in the previous 7 days;
* Are currently participating in an asthma-related pharmaceutical study or intervention study or has participated in another asthma-related pharmaceutical study or intervention study in the previous 4 weeks prior to recruitment;
* Are currently requiring greater than fluticasone 500 mcg bid plus long-acting beta agonist (LABA) 1 puff twice daily or its equivalent and\or individuals using oral corticosteroids daily or every other day at Visit 0.

Participants who meet any of the following criteria are not eligible for enrollment and may not be reassessed. Participants are ineligible if they:

* Have any medical illnesses that in the opinion of the investigators would a.) increase the risk the participant would incur by participating in the study, b.) interfere with the measured outcomes of the study, or c.) interfere with the performance of the study procedures. Examples of such diseases are: phenylketonuria, cystic fibrosis, bronchiectasis, Type 1 diabetes, hemophilia, Von Willebrands disease, sickle cell disease, cerebral palsy, rheumatoid arthritis, lupus, psoriasis, hyperimmunoglobulin E syndrome, parasite infections, Wiskott-Aldrich syndrome, or allergic bronchopulmonary aspergillosis.
* Have concurrent medical problems that would require systemic corticosteroids (other than for treatment of an asthma exacerbation) or other immunomodulators during the study;
* Currently have diagnosed cancer, are currently being investigated for possible cancer, or have a history of cancer;
* Have plans to move from the area during the study period;
* Do not primarily speak English (or Spanish at clinical sites with Spanish speaking staff);
* Have a primary caretaker who does not speak English (or Spanish at clinical sites with Spanish-speaking staff; not applicable if participant is able to provide consent);
* Are a foster child;
* Will not allow the study clinician to manage their disease for the duration of the study or are not willing to change their asthma medications to follow the protocol;
* Are not able to perform pulmonary function tests;
* Have known hypersensitivity to any of the medications that will be used for the treatment of asthma;
* Have had a life-threatening asthma exacerbation in the last 2 years requiring intubation, mechanical ventilation, or resulting in a hypoxic seizure.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The MUPPITS study will enroll inner-city children 6-17 years of age with difficult-to-control, exacerbation-prone asthma. Approximately 150 children will be enrolled and followed prospectively.
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2015-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Gene expression of nasal lavage RNA samples. | 6 month
  Gene expression will be measured by whole transcriptome RNA sequencing.

SECONDARY OUTCOMES:
Gene expression of whole blood RNA samples | 6 month
  Gene expression will be measured by whole transcriptome RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Jackson, MD, Principal Investigator — University of Wisconsin, Madison; Matthew C Altman, MD, MPhil, Study Chair — Benaroya Research Institute
Locations (9):
- United States (9):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann and Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston University School of Medicine, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: History, project and sites of the Inner-city Asthma Consortium (ICAC) — https://www.niaid.nih.gov/clinical-trials/inner-city-asthma-consortium
- See also: Information: National Asthma Education and Prevention Program (NAEPP) — http://www.nhlbi.nih.gov/about/org/naepp